CLINICAL TRIAL: NCT02449772
Title: Evaluation of ED Triage of Adult Patients With Alcohol Abuse
Brief Title: Emergency Department (ED) Triage of Alcohol Abuse
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Olivier T. Rutschmann, MD, MPH, University Hospital, Geneva
Other Study IDs: CER-14083R
Record Dates: First submitted 2015-04-28; First posted 2015-05-20 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Alcoholic Intoxication
Keywords: N04.452.442.422.336
MeSH Terms: conditions — Alcoholic Intoxication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Retrospective study of adult patients (> 16 y) admitted to Geneva University Hospitals with alcohol abuse. Triage criteria will be reviewed. Patients characteristics and patient flow in the ED will be described.

DETAILED DESCRIPTION:
A retrospective analysis of triage notes and electronic medical records will be performed in order to identify how triage evaluation is performed accordingly to the Swiss Emergency Triage Scale criteria. The proportion of patients leaving without being seen will be computed. Caracteristics of these patients will be compared to patients with medical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Triage code = alcohol abuse
* > 16 y

Exclusion Criteria:

* No alcohol abuse identified at triage
* < 16 y

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all adult patients admitted during one year in the ED for alcoholic abuse
Sampling Method: Non-Probability Sample
Enrollment: 775 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Triage questions asked | participants will be followed for the duration of emergency department stay, an expected average of 12 hours
  Number of questions asked at triage and proportion of patients with the full set of triage questions asked
Triage vital signs measured | participants will be followed for the duration of emergency department stay, an expected average of 12 hours
  Number of vital signs measured at triage and proportion of patients with the full set of triage vital signs measured
Number of undertriage | participants will be followed for the duration of emergency department stay, an expected average of 12 hours
  Number of patients with level 3 emergency levels attributed instead of level 2
Number of mistriage | participants will be followed for the duration of emergency department stay, an expected average of 12 hours
  Number of patients with erroneous triage reason attributed

SECONDARY OUTCOMES:
% of patients leaving without being seen | participants will be followed for the duration of emergency department stay, an expected average of 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Olivier T Rutschmann, MD, MPH, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, ED, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Dugas S, Favrod-Coune T, Poletti PA, Huwyler T, Richard-Lepouriel H, Simon J, Sarasin FP, Rutschmann OT. Pitfalls in the triage and evaluation of patients with suspected acute ethanol intoxication in an emergency department. Intern Emerg Med. 2019 Apr;14(3):467-473. doi: 10.1007/s11739-018-2007-7. Epub 2018 Dec 14. PMID 30552626